CLINICAL TRIAL: NCT01542905
Title: Effects of Korean Red Ginseng on Stress Relief and Cognitive and Mental Function Enhancement Using Neuroimaging: Double-Blind, Randomized, Placebo-Controlled Clinical Trial
Brief Title: Stress Relief Effect of Korean Red Ginseng
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In Kyoon Lyoo, MD, PhD, MMS, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KG2010
Record Dates: First submitted 2012-02-26; First posted 2012-03-02 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Stress Relief
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Korean Red Ginseng (Experimental)
  Interventions: Dietary Supplement: Korean Red Ginseng
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Korean Red Ginseng — Korean Red Ginseng Capsule (1g/day) for 8 Weeks
  Arms: Korean Red Ginseng
Other: Placebo — Placebo Capsule (1g/day) for 8 Weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine clinical and neuropsychiatric effects of Korean Red Ginseng and examine changes in brain structure, function and metabolites. A total of 60 healthy volunteers will be recruited and will be assigned to either Korean Red Ginseng group or placebo group. Individuals will be examined through clinical assessment, neuropsychological function tests and neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18~65

Exclusion Criteria:

* Current or past medical history, medical illnesses that are detected during clinical and physical evaluations
* Current Axis 1 diagnosis or past history of schizophrenia, bipolar, or psychotic disorders assessed by SCID-IV
* Current diagnosis of substance abuse assessed by SCID-IV
* Taking or have taken psychiatric medication in the past 2 months
* Head trauma accompanied by loss of consciousness or seizure
* IQ 80 or below
* Planning pregnancy, currently pregnant, or breastfeeding
* Claustrophobia or other fMRI incompatible factors such as pace makers
* Taking drugs, including over the counter drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Stress Scores at 8 Weeks | Baseline and 8 Weeks
Change from Baseline in Stress Scores at 4 Weeks | Baseline and 4 Weeks
Change from Baseline in Stress Scores at 1 Week | Baseline and 1 Week
Change from Baseline in Neurocognitive Function at 8 Weeks | Baseline and 8 Weeks
Change from Baseline in Brain Function, Chemistry, and Structure Measured Using Magnetic Resonance Imaging at 8 Weeks | Baseline and 8 Weeks

SECONDARY OUTCOMES:
Change in Fatigue Scores at 8 Weeks | Baseline and 8 Weeks
Change in Fatigue Scores at 4 Weeks | Baseline and 4 Weeks
Change in Fatigue Scores at 1 Week | Baseline and 1 Week
Change in Depressive Scores at 8 Weeks | Baseline and 8 Weeks
Change in Depressive Scores at 4 Weeks | Baseline and 4 Weeks
Change in Depressive Scores at 1 Week | Baseline and 1 Week
Change in Anxiety Scores at 8 Weeks | Baseline and 8 Weeks
Change in Anxiety Scores at 4 Weeks | Baseline and 4 Weeks
Change in Anxiety Scores at 1 Week | Baseline and 1 Week
Number of Participants Who Experienced Adverse Events | Week 1
Number of Participants Who Experienced Adverse Events | Week 4
Number of Participants Who Experienced Adverse Events | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: In Kyoon Lyoo, MD, PhD, MMS, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea